CLINICAL TRIAL: NCT01367951
Title: A Multi Centered Randomized Controlled Trial of Operative Versus Non-operative Treatment of Acute, Unstable Chest Wall Injuries
Brief Title: Treatment of Acute, Unstable Chest Wall Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Hamilton Health Sciences Corporation (Other); Vancouver General Hospital (Other); Eastern Health (Other); The Ottawa Hospital (Other); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unstable chest wall injuries
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Blunt Injury of Thorax; Flail Chest; Chest Wall Injury Trauma; Rib Fracture
Keywords: unstable chest injury; flail chest; chest wall injury; rib fracture
MeSH Terms: conditions — Flail Chest; Rib Fractures | interventions — Surgical Fixation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical fixation (Experimental): * The fractures will be reduced and stabilized by use of plates and screws
  * Attempt will be made to stabilize ribs 3-7, as these are surgically accessible and most important in maintaining integrity of the chest cavity.
  * Goal is not to fix all the fractures, but to fix sufficient fractures to create an internal splint and allow chest wall motion to occur as a unit. In case of fibs fractured at numerous locations, as many fragments will be reduced and stabilized as necessary to ensure movement as a unit.
  * Chest tube(s) will be placed at the discretion of the treating surgeon in patients with pre-operative or intra-operative violation of the pleural cavity (ie pre-op pneumothorax/haemothorax, iatrogenic pleural injury). No post-operative drains will be inserted.
  Interventions: Procedure: Surgical fixation
- non-operative (No Intervention): 1. Mechanical ventilation: Patients in respiratory distress will receive endotracheal intubation, and placed on mechanical ventilation. PEEP will be utilized as needed, at the discretion of the ICU and respiratory therapy team.
  2. Other conservative means/Pulmonary toilet:Patients will receive aggressive pulmonary toilet (suctioning of ET tube as needed), chest physiotherapy (as per standard local protocol), and will have the head of the bed elevated to 30° unless contraindicated (ie unstable C-spine injury).
  3. Pain control:Epidural catheters, intercostal nerve block, PCA, IV/PO pain medication

INTERVENTIONS:
Procedure: Surgical fixation — * The fractures will be reduced and stabilized by use of plates and screws
  * Attempt will be made to stabilize ribs 3-7, as these are surgically accessible and most important in maintaining integrity of the chest cavity.
  * Goal is not to fix all the fractures, but to fix sufficient fractures to create an internal splint and allow chest wall motion to occur as a unit. In case of fibs fractured at numerous locations, as many fragments will be reduced and stabilized as necessary to ensure movement as a unit.
  * Chest tube(s) will be placed at the discretion of the treating surgeon in patients with pre-operative or intra-operative violation of the pleural cavity (ie pre-op pneumothorax/haemothorax, iatrogenic pleural injury). No post-operative drains will be inserted.
  Arms: Surgical fixation

SUMMARY:
Unstable chest injuries are common in poly trauma patients. They can lead to severe pulmonary restriction, loss of lung volume, difficulty with ventilation and can render the patient to require intubation and mechanical ventilation. Traditionally these injuries have been treated non-operatively, however in the past decade there has been numerous studies suggesting improved outcomes with surgical fixation. Surgical fixation can significantly decrease time spent in ICU as well as day on mechanical ventilation. The investigators aim is to conduct a randomized control trial of these injuries, to compare non-operative treatment with surgical fixation. The investigators' hypothesis is that surgically treated patient will have significantly improved outcomes compared to those treated non-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Age >16 or skeletal maturity
* Meeting one of the two indication for surgical fixation of chest wall injury:

  1. Flail chest, defined as follows:

     * 3 unilateral segmental rib fractures; OR
     * 3 bilateral rib fractures; OR
     * 3 unilateral fractures combined with sternum fracture/dissociation Note: at least 3 of the rib fractures involved in the flail segment must demonstrate displacement.
  2. Severe deformity of the chest wall (Diagnosed by CT scan). Defined as follows:

     * Severe (100%) displacement of 3 or more ribs OR
     * Marked loss thoracic volume/caved in chest (>25% volume loss in involved lobe(s)); OR
     * Overriding of 3 or more rib fractures (by minimum 15mm each); OR
     * Two or more rib fractures associated with intra-parenchymal injury - ie ribs in the lung, in the parenchyma

Exclusion Criteria:

* Anatomic location of rib fractures are not amenable to surgical fixation (eg fractures directly adjacent to spinal column)
* Rib fractures primarily involving floating ribs (ribs 10-12)
* Home Oxygen (O2) requirement
* Other significant injuries that may require long term intubation:
* Severe pulmonary contusion (Defined as PaO2/FIO2 ratio <200 with radiological evidence of pulmonary infiltrates WITHIN 24 hours of THORACIC TRAUMA)
* Severe head injury/Traumatic brain injury - (GCS ≤ 8 at 48 hrs post injury. If unable to assess full GCS due to intubation or other causes, GCS motor ≤4 at 48 hrs post injury)
* Upper airway injury requiring long term intubation and mechanical ventilation (e.g. tracheal disruption)
* Acute quadriplegia/quadraparesis
* Head and neck burn injuries, or inhalation burn injuries
* Dementia or other inability to complete follow-up questionnaires
* Medically unstable for OR (e.g. haemodynamic instability, acidosis, coagulopathy, etc.)* or unlikely to survive 1 year follow-up, in the opinion of the attending physician
* Lack of informed consent from patient or substitute decision maker
* Randomization > 72 hours from injury
* ORIF > 96 hours from injury (if randomized to surgical fixation group)
* Age > 85

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2011-07; Primary Completion 2018-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days (VFD) | 28 Days
  To compare early surgical fixation versus conventional, non-surgical treatment of unstable chest injuries on the basis of our primary outcome measure of days spent free from a mechanical ventilator in the first 28 days following injury.

SECONDARY OUTCOMES:
Number of days in the Intensive Care Unit (ICU) | 12 months
  The total number of days in ICU will be calculated over the 12 months period post injury. If no ICU stay is needed the total days in ICU will be 0.
Amount of pain medication administration, converted to oral morphine equivalence | 4 weeks
  The total daily pain medication administration will be calculated, and converted to daily oral (PO) morphine equivalence.
Rate of Pneumonia | 12 months
  The number of times patient is diagnosed with pneumonia over 12 months post injury
Pulmonary function assessment | 12 months
  spirometry measurement of total lung capacity (TLC), forced vital capacity (FVC) and forced expiratory volume at 1 second (FEV1), measured at 3 months and at 12 months post injury
Rate of return to work | 12 months
  to assess if patient has returned to work at 12 months, and at what capacity
assessment of functional health and well being | 12 months
  Using SF-36 questionnaire we will assess the patient's well-being and functional health

CONTACTS AND LOCATIONS:
Overall Officials: Michael D McKee, MD, FRCS(C), Principal Investigator — St. Michael's Hospital, University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dehghan N, Nauth A, Schemitsch E, Vicente M, Jenkinson R, Kreder H, McKee M; Canadian Orthopaedic Trauma Society and the Unstable Chest Wall RCT Study Investigators. Operative vs Nonoperative Treatment of Acute Unstable Chest Wall Injuries: A Randomized Clinical Trial. JAMA Surg. 2022 Nov 1;157(11):983-990. doi: 10.1001/jamasurg.2022.4299. PMID 36129720